CLINICAL TRIAL: NCT00706160
Title: Noninvasive Language Mapping in Patients With Localization-Related Epilepsy
Brief Title: Language Mapping in Patients With Epilepsy
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080161; 08-N-0161
Record Dates: First submitted 2008-06-26; First posted 2008-06-27 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-04-04

CONDITIONS: Epilepsy; Epilepsy, Temporal Lobe; Partial Epilepsy
Keywords: Epilepsy; Language; fMRI; Magnetoencephalogram; Temporal Lobe Epilepsy; Partial Epilepsy; Healthy Volunteer; HV
MeSH Terms: conditions — Epilepsy; Epilepsy, Temporal Lobe; Epilepsies, Partial; Language

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will examine how certain language skills, such as naming objects, understanding spoken language and reading are organized in the brain and how they are affected by seizures.

People with epilepsy who are considering surgery and healthy volunteers who are right-handed and between the ages of 7 and 55 may be eligible for this study. Participants undergo the following procedures twice, and, in some cases, possibly three times, in two or three visits of 2 to 4 hours each.

Neuropsychological tests: Testing includes questionnaires, pen-and-pencil or computerized tests and motor tasks.

Structural MRI: This procedure uses a strong magnetic field and radio waves to obtain pictures of brain structure. During the test, the subject lies in the scanner (a metal cylinder surrounded by a magnetic field) for about 90 minutes, wearing earmuffs to muffle knocking noises the machine makes. Subjects may be asked to lie still for up to 10 minutes at a time.

Functional MRI: This procedure is similar to structural MRI, except a coil is placed over the head and the subject performs simple tasks during the procedure. The pictures obtained show what parts of the brain are being used to perform the task. The test lasts about 60 minutes, with subjects asked to lie still for up to 10 minutes at a time.

Magnetoencephalography (MEG) and electroencephalography (EEG): For MEG, the subject sits in an MEG recording room with a cone containing magnetic field detectors lowered onto his or her head. Very small magnetic changes produced by the activity of the brain are recorded while the subject sits quietly or performs a research task. An EEG recording of the electrical activity of the brain is done at the same time as the MEG.

...

DETAILED DESCRIPTION:
Objective: This protocol will test the hypothesis that successful left hemisphere epilepsy surgery for children and adults improves abnormalities in the functional anatomy of language that may be associated with uncontrolled localization-related seizures. We will use an established modality, functional magnetic resonance imaging (fMRI), which has been used extensively for evaluation of patients with epilepsy, as our primary outcome measure, and an emerging modality, magnetoencephalography (MEG), as a secondary measure. We will explore methods of MEG data analysis for comparison with fMRI results.

Study Population:

150 patients with localization-related epilepsy who are surgical candidates and 50 healthy volunteers.

Design: This is a non-invasive imaging study that will employ a test battery including standard neuropsychological tests, structural MRI, fMRI, and a 275-channel whole-head MEG recording, for evaluation of the functional anatomy of language. The test battery will be performed pre-operatively and at 12 months after surgery.

Main outcome measure: Measurement of the "laterality index" comparing left and right hemisphere regional activation on fMRI before and after surgery, in patients after left sided or right-sided surgery, and healthy controls.

Secondary outcome measure: Measurement of the "laterality index" comparing left and right hemisphere regional activation on MEG before and after surgery.

ELIGIBILITY:
* INCLUSION CRITERIA FOR PATIENTS:

  1. Age 7-55
  2. Documentation of localization-related epilepsy based on clinical, neuropsychological and imaging criteria
  3. Failure of seizures to respond to adequate therapy with at least two standard antiepileptic drugs
  4. Willingness to be considered for surgery
  5. Fluency in English. Non-native speakers may be included if their fluency is equivalent to that of a native speaker.

INCLUSION CRITERIA FOR HEALTHY VOLUNTEERS:

1. Age 7-55
2. Willingness to participate in and complete the study
3. Right-handedness assessed by the Edinburg handedness inventory
4. Fluency in English

EXCLUSION CRITERIA FOR PATIENTS:

1. Contra-indications to MRI studies (such as pacemakers, cochlear devices, surgical clips etc. metallic implants, orthopedic pins, shrapnel, permanent eyeliner, vagus nerve stimulator)
2. Claustrophobia or anxiety disorders exacerbated by the MRI scanner
3. People with neurological or psychiatric disease or taking medications that would affect fMRI and MEG language studies
4. Pregnancy. All females of child bearing potential must have a negative test prior to MRI scanning
5. Patients on phenobarbital or chronic benzodiazepines

EXCLUSION CRITERIA FOR HEALTHY VOLUNTEERS:

1. Contra-indications MRI studies (metallic implants, recent orthopedic pins, cochlear implants, surgical clips, cardiac pacemakers and defibrillation devices, shrapnel, permanent eyeliner, vagus nerve stimulator)
2. Any medical condition or chronic medication that might affect fMRI or MEG language activation by affecting cerebral structure or function, such as diabetes, hypertension, antihypertensive medications, psychotropic agents.
3. Pregnancy. All females of child bearing potential must have a negative test prior to MRI scanning.

Ages: 7 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 153 (Actual)
Dates: Start 2008-06-13; Study Completion 2013-04-04

PRIMARY OUTCOMES:
Change in asymmetry index of fMRI after surgery.

SECONDARY OUTCOMES:
Changes in asymmetry index on MEG after surgery and seizure control after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: William H Theodore, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Berl MM, Balsamo LM, Xu B, Moore EN, Weinstein SL, Conry JA, Pearl PL, Sachs BC, Grandin CB, Frattali C, Ritter FJ, Sato S, Theodore WH, Gaillard WD. Seizure focus affects regional language networks assessed by fMRI. Neurology. 2005 Nov 22;65(10):1604-11. doi: 10.1212/01.wnl.0000184502.06647.28. PMID 16301489
- [Background] Binder JR, Swanson SJ, Hammeke TA, Morris GL, Mueller WM, Fischer M, Benbadis S, Frost JA, Rao SM, Haughton VM. Determination of language dominance using functional MRI: a comparison with the Wada test. Neurology. 1996 Apr;46(4):978-84. doi: 10.1212/wnl.46.4.978. PMID 8780076
- [Background] Brookes MJ, Vrba J, Robinson SE, Stevenson CM, Peters AM, Barnes GR, Hillebrand A, Morris PG. Optimising experimental design for MEG beamformer imaging. Neuroimage. 2008 Feb 15;39(4):1788-802. doi: 10.1016/j.neuroimage.2007.09.050. Epub 2007 Oct 10. PMID 18155612